CLINICAL TRIAL: NCT03786718
Title: Usability of Diabetes Dashboard Embedded Within a Patient Web Portal: A Prospective Longitudinal Study
Brief Title: Usability of Diabetes Dashboard Embedded Within a Patient Web Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 181727; 5K23DK106511 (NIH)
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Patient Web Portals; Usability; Health Information Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients have access to a patient web portal with the Patient-facing Diabetes Dashboard activated.
  Interventions: Other: Patient-facing Diabetes Dashboard

INTERVENTIONS:
Other: Patient-facing Diabetes Dashboard — The Patient-facing Diabetes Dashboard is embedded within a patient web portal and includes graphics to visualize and summarize patients' health data, incorporates motivational strategies (e.g., social comparisons and gamification), provides literacy level appropriate educational resources, and contains secure-messaging capability.

SUMMARY:
The purpose of this study is to conduct a prospective, longitudinal study to evaluate the usability of a patient-facing diabetes dashboard delivered via an established patient web portal.

DETAILED DESCRIPTION:
Up to 70 adult patients with type 2 diabetes mellitus will be enrolled and given access to a diabetes dashboard within an existing patient web portal. Patients will be invited by mail (or email) to be screened for enrollment in the study. Patients may also respond at a study flyer and contact the study team to be screened for enrollment. Eligible and interested patients will be emailed a link to a secure study website where they will complete a web consent form. After enrollment, participants will complete a baseline web-based questionnaire. After completing the enrollment questionnaire, they will be provided access to the diabetes dashboard within the patient web portal for one month. After one month, participants will receive an additional follow-up (final) questionnaire to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Currently being treated with at least one antihyperglycemic medication
* Able to speak and read in English
* Have reliable access to a computer with internet access
* Existing My Health at Vanderbilt (i.e., patient portal) account

Exclusion Criteria:

* Living in long term care facilities
* Known cognitive deficits
* Severe visual or hearing impairment
* Unintelligible speech (e.g., dysarthria)
* Currently participating in another diabetes-related research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- William Martinez, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 69 enrolled participants, 67 completed the baseline questionnaire and were with given access to the intervention. Two participants never completed the baseline questionnaire despite reminders and therefore did not receive access to the intervention and were withdrawn.
Groups:
- Intervention: Patients have access to a patient web portal with the Patient-facing Diabetes Dashboard activated.
  Patient-facing Diabetes Dashboard: The Patient-facing Diabetes Dashboard (also known as My Diabetes Care) is embedded within a patient web portal and includes graphics to visualize and summarize patients' health data, incorporates motivational strategies (e.g., social comparisons), provides literacy level appropriate educational resources, and contains secure-messaging capability.
Period: Overall Study
Arm/Group | Intervention
Started | 67
Completed | 60
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Did not use the intervention | 2
Not completed — diagnosis changed from type 2 to type 1 | 1

BASELINE CHARACTERISTICS:
Population: 67 participants were provided access to the intervention, however, analysis was limited to 60 participants who completed the study (i.e., used the intervention and submitted both pre- and post-study questionnaires).
Arm/Group | Intervention
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 41
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 60
Education [Count of Participants; unit: Participants]
  High school/GED | 5
  Some college/technical school | 24
  College degree | 19
  Graduate or professional degree | 12
Health Literacy [Count of Participants; unit: Participants] — Health literacy was assessed using a validated one-item screener that asked respondents to rate their confidence independently filling out medical forms on a scale ranging from 'extremely' to 'not at all' confident. Consistent with prior studies, we categorized participants noting any lack of confidence filling out medical forms as having limited health literacy.
  Participants
    Adequate | 31
    Limited | 29
eHealth Literacy [Mean (Standard Deviation); unit: units on a scale] — eHealth refers to healthcare services provided electronically via the Internet. eHealth Literacy refers to the knowledge, comfort, and perceived skill at finding, evaluating, and applying electronic health information to health problems. eHealth Literacy was assessed by the eHEALS scale which contains 8 items, measured with a 5-point Likert scale with response options ranging from "strongly disagree=1" to "strongly agree=5." Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy. Population: One participant did not complete the eHEALS scale
  units on a scale
    number analyzed (Participants) | 59
    (all) | 31.5 (5.2)
Patient Portal Usage [Count of Participants; unit: Participants]
  Weekly | 26
  Monthly | 29
  Other | 5
Computer and Smartphone Usage [Number; unit: participants] — Participants could select more than one so totals may exceed 100%.
  participants
    Desktop | 50
    Tablet | 40
    Smartphone | 52
Hemoglobin A1c [Mean (Standard Deviation); unit: %] — Population: Two participants were missing hemoglobin A1C data.
  %
    number analyzed (Participants) | 58
    (all) | 7.5 (1.6)
Insulin Use [Count of Participants; unit: Participants]
  Yes | 24
  No | 36
Time with diagnosis of diabetes [Mean (Standard Deviation); unit: years] | 13.1 (10.0)
Comorbidities [Number; unit: participants] — Number of participants with comorbid hyperlipidemia and/or hypertension
  participants
    Hyperlipidemia | 47
    Hypertension | 51

OUTCOME MEASURES:

1. Primary Outcome: Usability
Description: The System Usability Scale (SUS) will be administered to all study participants at one month follow-up (T1). The SUS is a validated measure of usability. The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). A score of above 68 indicative of "above average" usability.
Time Frame: one month follow-up (T1)
Population: All 60 participants that completed the study (i.e., used the intervention and complete pre- and post-questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 60
score on a scale | 78.8 [72.5 to 87.5]
Statistical Analysis 1: Comparison: Intervention; Due to nonnormality, we used nonparametric tests to analyze the data. This analysis is a one sample median test of participants' median SUS score compared to the threshold score of 68 indicative of 'above average' usability; Test type: Other; p < 0.001, One sample median test

2. Primary Outcome: User Experience - Quantitative
Description: User experience will be assessed by study-specific survey items administered to all study participants at the end of the study period (T1). The survey items will inquire about participants' perspectives on particular features of the Patient-facing Diabetes Dashboard. Participants were asked to indicate which features, if any: (1) they found useful for managing their diabetes and which features, (2) improved their understanding of their diabetes health data, and (3) should be removed. In addition, participants indicated whether they intended to use the dashboard going forward if it remained available.
Time Frame: one month follow-up (T1)
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
participants
  Star Status Indicator - useful | 19
  Hover Over Info Icons - useful | 26
  Goal, Caution, and Warning Ranges - useful | 46
  Patients Like Me Data - useful | 40
  Literacy Sensitive Education Links - useful | 40
  Diabetes Online Community - useful | 22
  Star Status Indicator - understanding | 18
  Hover Over Info Icons - understanding | 31
  Goal, Caution, and Warning Ranges - understanding | 39
  Literacy Sensitive Education Links - understanding | 39
  Diabetes Online Community - understanding | 15
  Star Status Indicator - removed | 4
  Hover Over Info Icons - removed | 0
  Goal, Caution, and Warning Ranges - removed | 2
  Patients Like Me Data - removed | 4
  Literacy Sensitive Education Links - removed | 0
  Diabetes Online Community - removed | 1
  Intend to use going forward | 60

3. Primary Outcome: User Experience - Qualitative
Description: At the end of the study period (T1), a subset of study participants will be invited to complete a semi-structured interview to provide a deeper understanding of their experience using the dashboard.
Time Frame: one month follow-up (T1)
Population: participants that participated in a semi-structured interview
Measure: Number; unit: areas for improvement identified
Arm/Group | Intervention
Number analyzed (Participants) | 14
areas for improvement identified | 5

4. Secondary Outcome: System Usage Data
Description: This is a composite outcome measure of participants' self-reported total number of diabetes dashboard visits, total duration of dashboard use, use of embedded educational links, utilization of embedded functionality to secure message healthcare team member(s), and use of an embedded link to American Diabetes Association Online Community and will be queried at the end of the study period (T1).
Time Frame: one month follow-up (T1)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
Participants
  Total number of visits: 1-2 | 12
  Total number of visits: 3-4 | 27
  Total number of visits: 5-6 | 12
  Total number of visits: 7+ | 9
  Total minutes spent: <5 minutes | 4
  Total minutes spent: 5-9 minutes | 7
  Total minutes spent: 10-14 minutes | 19
  Total minutes spent: 15+ minutes | 30
  Used literacy sensitive education links | 51
  Used secure messaging | 10
  Used diabetes online community | 16
  Used info icon with explanation of health measure | 49

5. Secondary Outcome: Change in Diabetes Knowledge
Description: The Short Diabetes Knowledge Instrument (SDKI) was used to measure diabetes knowledge including diabetes diet, symptoms of hypoglycemia, foot care and importance of physical activity. The SDKI is a 13-item scale with scores ranging from 0 to 13 representing number of items answered correctly. The Short Diabetes Knowledge Instrument (SDKI) will be administered to all study patients at enrollment (T0) and one month follow-up (T1).
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: Missing data for one participant
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 59
score on a scale
  enrollment (T0) | 11.0 [10 to 12]
  one month follow-up (T1) | 11.0 [10 to 12]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.77, Wilcoxon Signed Rank Sum test

6. Secondary Outcome: Change in Diabetes Self-Care
Description: Diabetes self-care will be measured using the Summary of Diabetes Self-Care Activities (SDSCA), an 11-item questionnaire of diabetes self-management that assess the following six aspects of the diabetes regimen: general diet (2 items), specific diet (2 items), exercise (2 items), blood-glucose testing (2 items), foot care (2 items), and smoking (1 items). Item responses use the metric "days per week" except for a single item about smoking status which is yes or no. Each of the five aspects (excluding smoking) is assigned a mean score based on number of days per week. The Summary of Diabetes Self-Care Activities (SDSCA) will be administered to all study patients at enrollment (T0) and one month follow-up (T1).
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: The overall number of participants analyzed for two blood-glucose testing items was 50, because 10 participants that do not test their blood sugar were excluded from those two items. Overall number of participants analyzed was 60 for the the other five aspects/sub-scales.
Measure: Median (Inter-Quartile Range); unit: days per week
Arm/Group | Intervention
Number analyzed (Participants) | 60
days per week
  general diet at enrollment (T0) | 4.0 [2.8 to 5.0]
  general diet at one month follow-up (T1) | 4.0 [3.5 to 5.0]
  specific diet at enrollment (T0) | 3.5 [2.0 to 5.0]
  specific diet at one month follow-up (T1) | 4.0 [2.5 to 5.0]
  exercise at enrollment (T0) | 2.5 [0.5 to 3.8]
  exercise at one month follow-up (T1) | 2.3 [1.3 to 4.0]
  blood-glucose testing at enrollment (T0): number analyzed (Participants) | 50
  blood-glucose testing at enrollment (T0) | 5.3 [3.0 to 7.0]
  blood-glucose testing at one month follow-up (T1): number analyzed (Participants) | 50
  blood-glucose testing at one month follow-up (T1) | 6.0 [3.0 to 7.0]
  foot care at enrollment (T0) | 3.5 [1.0 to 4.8]
  foot care at one month follow-up (T1) | 3.0 [1.0 to 5.0]
Statistical Analysis 1: Comparison: Intervention; Analysis for pre-post change in General Diet sub-scale score; Test type: Other; p = 0.02, Wilcoxon Signed Rank Sum test
Statistical Analysis 2: Comparison: Intervention; Analysis for pre-post change in Specific Diet sub-scale score; Test type: Other; p = 0.13, Wilcoxon Signed Rank Sum test
Statistical Analysis 3: Comparison: Intervention; Analysis for pre-post change in Exercise sub-scale score; Test type: Other; p = 0.35, Wilcoxon Signed Rank Sum test
Statistical Analysis 4: Comparison: Intervention; Analysis for pre-post change in Blood-glucose Testing sub-scale score; Test type: Other; p = 0.67, Wilcoxon Signed Rank Sum test
Statistical Analysis 5: Comparison: Intervention; Analysis for pre-post change in Foot Care sub-scale score; Test type: Other; p = 0.65, Wilcoxon Signed Rank Sum test

7. Secondary Outcome: Change in Diabetes Self-Efficacy
Description: The Perceived Diabetes Self-Management Scale (PDSMS) is a valid measure of diabetes self-efficacy. The PDSMS will be administered to all study participants at enrollment (T0) and one month follow-up (T1). Eight items are scored on a five-point Likert scale. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: One participant had missing data.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 59
score on a scale
  enrollment (T0) | 26.0 [23.0 to 30.0]
  one month follow-up (T1) | 29.0 [25.0 to 32.0]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.001, Wilcoxon Signed Rank Sum test

8. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. The PAID-5 will be administered to all study participants at enrollment (T0) and one month follow-up (T1). Total scores on the PAID-5 can range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress.
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: Missing data for one participant.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 59
score on a scale
  enrollment (T0) | 5.0 [2.0 to 9.0]
  one month follow-up (T1) | 5.0 [2.0 to 9.0]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.86, Wilcoxon Signed Rank Sum test

9. Secondary Outcome: Change in Knowledge of Diabetes Measures
Description: Unique study specific items to assess participants' knowledge of measures of diabetes health status (e.g., Hemoglobin A1C) will be administered to all study participants at enrollment (T0) and one month follow-up (T1).
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: As noted in the outcome measure data table below, the number analyzed for some items is less than 60 due to missing data.
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
participants
  Identify definition of A1c at T0: number analyzed (Participants) | 58
  Identify definition of A1c at T0 | 40
  Identify definition of A1c at T1: number analyzed (Participants) | 58
  Identify definition of A1c at T1 | 45
  Identify goal range for A1c at T0: number analyzed (Participants) | 59
  Identify goal range for A1c at T0 | 50
  Identify goal range for A1c at T1: number analyzed (Participants) | 59
  Identify goal range for A1c at T1 | 50
  Identify definition of blood pressure at T0: number analyzed (Participants) | 59
  Identify definition of blood pressure at T0 | 43
  Identify definition of blood pressure at T1: number analyzed (Participants) | 59
  Identify definition of blood pressure at T1 | 46
  Identify goal range for blood pressure at T0: number analyzed (Participants) | 59
  Identify goal range for blood pressure at T0 | 17
  Identify goal range for blood pressure at T1: number analyzed (Participants) | 59
  Identify goal range for blood pressure at T1 | 28
  Identify definition of LDL cholesterol at T0: number analyzed (Participants) | 59
  Identify definition of LDL cholesterol at T0 | 22
  Identify definition of LDL cholesterol at T1: number analyzed (Participants) | 59
  Identify definition of LDL cholesterol at T1 | 25
  Identify goal range for LDL cholesterol at T0: number analyzed (Participants) | 58
  Identify goal range for LDL cholesterol at T0 | 15
  Identify goal range for LDL cholesterol at T1: number analyzed (Participants) | 58
  Identify goal range for LDL cholesterol at T1 | 31
  Identify definition of flu vaccine at T0 | 58
  Identify definition of flu vaccine at T1 | 59
  Identify frequency of flu vaccination at T0 | 58
  Identify frequency of flu vaccination at T1 | 59
Statistical Analysis 1: Comparison: Intervention; Analysis for pre-post change in knowledge of definition of A1C; Test type: Other; p = 0.30, McNemar
Statistical Analysis 2: Comparison: Intervention; Analysis for pre-post change in knowledge of goal range for hemoglobin A1c; Test type: Other; p = 1.00, McNemar
Statistical Analysis 3: Comparison: Intervention; Analysis for pre-post change in knowledge of definition of systolic blood pressure; Test type: Other; p = 0.63, McNemar
Statistical Analysis 4: Comparison: Intervention; Analysis of pre-post change in knowledge of goal range for systolic blood pressure; Test type: Other; p = 0.02, McNemar
Statistical Analysis 5: Comparison: Intervention; Analysis of pre-post change in knowledge of definition of LDL cholesterol; Test type: Other; p = 0.55, McNemar
Statistical Analysis 6: Comparison: Intervention; Analysis for pre-post change in knowledge of goal range for LDL cholesterol; Test type: Other; p = 0.0009, McNemar
Statistical Analysis 7: Comparison: Intervention; Analysis of pre-post change in knowledge of definition of flu vaccine; Test type: Other; p = 1.00, McNemar
Statistical Analysis 8: Comparison: Intervention; Analysis of pre-post change in knowledge of recommended frequency of flu vaccination; Test type: Other; p = 1.00, McNemar

10. Secondary Outcome: Change in Diabetes Understanding
Description: The Diabetes Care Profile (DCP) is a self-administered questionnaire that assesses the social and psychological factors related to diabetes and its treatment. The instrument includes sixteen scales. The Understanding Scale of the DCP contains 13 items that assesses respondents' perceived understanding of elements of diabetes self-care (e.g., diet for blood sugar control). We administered 9 of the 13 items to study participants, excluding items that referenced elements of self-management that are not covered in My Diabetes Care (e.g., pregnancy and diabetes). Respondents rate their understanding on a five-point Likert scale. The scale scores range from 1 to 5 and represents the average item score for the scale (∑ Q1-9/ Count of non-missing items). High scores indicate higher perceived understanding.
Time Frame: enrollment (T0) and one month follow-up (T1)
Population: Missing data for one participant
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 59
score on a scale
  enrollment (T0) | 3.4 [3.0 to 4.0]
  one month follow-up (T1) | 3.7 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.15, Wilcoxon Signed Rank Sum test

11. Secondary Outcome: Change in Attitudes
Description: Unique study specific survey items to assess participants' attitudes toward receiving social and goal-based comparison information regarding their diabetes health status will be administered to all study participants at enrollment (T0) and one month follow-up (T1).
Time Frame: enrollment (T0) and one month follow-up (T1)
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
participants
  Interested in social comparison info at T0 | 51
  Interested in social comparison info at T1 | 46
  Interested goal-based comparison info at T0 | 58
  Interested goal-based comparison info at T1 | 59
  Agree social comparison info is useful at T0 | 49
  Agree social comparison info is useful at T1 | 46
  Agree goal-based comparison info is useful at T0 | 59
  Agree goal-based comparison info is useful at T1 | 57
Statistical Analysis 1: Comparison: Intervention; Analysis of pre-post change in interest in information about how my diabetes health data compares to other patients like me (i.e., social comparison information); Test type: Other; p = 0.23, McNemar
Statistical Analysis 2: Comparison: Intervention; Analysis of pre-post change in interest in information about how their diabetes health data compares to the goal range (i.e., goal-based comparison information); Test type: Other; p = 1.00, McNemar
Statistical Analysis 3: Comparison: Intervention; Analysis of pre-post change in agreement with statement: 'Information about how my diabetes health data compares to other patients like me [social comparison information] is useful.'; Test type: Other; p = 0.51, McNemar
Statistical Analysis 4: Comparison: Intervention; Analysis of pre-post change in agreement with statement: 'Information about how my diabetes health data compares to the goals range [goal-based comparison information] is useful; Test type: Other; p = 0.63, McNemar

12. Secondary Outcome: Change in Patient Activation
Description: The Patient Activation Measure® (PAM-13) scale will be administered to all study participants at enrollment (T0) and one month follow-up (T1). The 13-item PAM® survey is a validated measure of patient activation (i.e., the knowledge, skills and confidence a person has in managing their own health and health care) and consists of 13 items. Each item uses a 4-point Likert-type scale of response options ranging from strongly disagree to strongly agree to elicit endorsement of a particular statement. PAM® survey item responses result in total raw scores ranging from 13 to 52, which we converted to the linear interval scale of patient activation scores, ranging from 0 (lowest activation) to 100 (highest activation).
Time Frame: enrollment (T0) and one month follow-up (T1)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 60
score on a scale
  enrollment (T0) | 64.3 [55.6 to 72.5]
  one month follow-up (T1) | 67.8 [60.6 to 75.0]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.01, Wilcoxon Signed Rank Sum test

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT03786718/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03786718/ICF_000.pdf